CLINICAL TRIAL: NCT06543706
Title: Metabolic Syndrome and Its Related Diseases in Healthcare Workers: Incidence, Prevalence, and Risk Factors
Brief Title: Metabolic Syndrome and Related Diseases in Healthcare Workers
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: K2557
Record Dates: First submitted 2024-06-06; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-06

CONDITIONS: Metabolic Syndrome X; Diabetes Mellitus Type 2; Hypertension; Hyperlipidemia; Obesity; Cardiovascular Diseases; Stroke
Keywords: metabolic syndrome; metabolic related diseases; medical workers
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Hypertension; Hyperlipidemias; Obesity; Cardiovascular Diseases; Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- the Metabolic Related Diseases in Medical Workers (MRDMW) cohort: The cohort includes all hospital employees who receive annual check-ups.

SUMMARY:
This study aims to investigate the incidence and prevalence of metabolic syndrome and metabolism-related diseases among healthcare workers, identify potential risk factors for these diseases, evaluate the control status of these conditions, and explore the significance of annual regular check-ups in improving metabolic-related health outcomes. All data for the study subjects are sourced from anonymized continuous records in hospital physical examinations and medical case files. The study does not involve any interventions. Upon obtaining the study data, researchers will use retrospective analysis methods to identify possible associations between risk factors and diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Healthcare workers who attend annual check-ups at Peking Union Medical College Hospital

Exclusion Criteria:

* Presence of metabolic syndrome, hypertension, diabetes, coronary heart disease, or stroke at the time of the first physical examination between 2012 and 2022
* Malignant neoplasm
* Uremia
* Liver failure
* Moderate to severe heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthcare workers who were working in the hospital, including those who have retired from the hospital
Sampling Method: Non-Probability Sample
Enrollment: 7432 (Actual)
Dates: Start 2022-11-18 (Actual); Primary Completion 2023-08-07 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
composite endpoint of cardiovascular and cerebrovascular diseases | through study completion, an average of 5 years
  The number of hospitalizations due to severe coronary heart disease, stroke, or sudden cardiac death. The outcome is determined if any of the first three discharge diagnoses include acute myocardial infarction, stroke, or sudden cardiac death, or if an emergency coronary stent placement or coronary artery bypass graft surgery is performed during hospitalization.

SECONDARY OUTCOMES:
new-onset metabolic syndrome | through study completion, an average of 5 years
  The number of individuals who did not meet the criteria for metabolic syndrome at the first examination but developed the syndrome later. The diagnostic criteria for metabolic syndrome involve meeting three or more of the following conditions:
  Abdominal obesity: waist circumference ≥90 (men) or ≥85 (women) cm. Hyperglycemia: fasting blood glucose ≥6.1 or 2-hour postprandial blood glucose ≥7.8 mmol/L or previously diagnosed diabetes. Hypertension: blood pressure ≥130/85 mmHg or previously diagnosed hypertension. Elevated triglycerides: fasting triglycerides ≥1.70 mmol/L or on lipid-lowering medication. Low fasting high-density lipoprotein cholesterol (HDL-C) <1.04 mmol/L.
  If waist circumference and HDL-C data are missing, abdominal obesity will be defined using the body mass index (BMI), calculated by dividing weight in kilograms by the square of height in meters (BMI ≥ 28.0 kg/m^2). Total cholesterol ≥ 5.17 mmol/L will be used as a substitute for the HDL-C indicator.

CONTACTS AND LOCATIONS:
Overall Officials: Tengda Xu, Principal Investigator — Department of Health, Peking Union Medical College Hospital
Locations (1):
- Tengda Xu, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Individual patient data (IPD) could be shared with other researchers after the publication of the study. However, the sharing should be permitted by the principal investigator from email. We do not have a web address for finding more information about the individual patient data (IPD) sharing plan. And we reject any data requests with commercial intentions.

REFERENCES:
- [Result] Strauss M, Lavie CJ, Lippi G, Brzek A, Vollenberg R, Sanchis-Gomar F, Leischik R. A systematic review of prevalence of metabolic syndrome in occupational groups - Does occupation matter in the global epidemic of metabolic syndrome? Prog Cardiovasc Dis. 2022 Nov-Dec;75:69-77. doi: 10.1016/j.pcad.2022.09.003. Epub 2022 Sep 23. PMID 36162483
- [Result] Liu J, Liu Q, Li Z, Du J, Wang C, Gao Y, Wei Z, Wang J, Shi Y, Su J, Liu Y, Wang P, Xie C, Li G, Shao B, Zhang L. Prevalence of Metabolic Syndrome and Risk Factors Among Chinese Adults: Results from a Population-Based Study - Beijing, China, 2017-2018. China CDC Wkly. 2022 Jul 22;4(29):640-645. doi: 10.46234/ccdcw2022.138. PMID 35919823
- [Result] Xi B, He D, Hu Y, Zhou D. Prevalence of metabolic syndrome and its influencing factors among the Chinese adults: the China Health and Nutrition Survey in 2009. Prev Med. 2013 Dec;57(6):867-71. doi: 10.1016/j.ypmed.2013.09.023. Epub 2013 Oct 5. PMID 24103567